CLINICAL TRIAL: NCT05379465
Title: The Impact of the COVID-19 Pandemic on the Career Choice of Medicine: A Cross-Sectional Study Amongst Pre-Medical Students in Pakistan
Brief Title: The Impact of the COVID-19 Pandemic on the Career Choice of Medicine
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sarah Nadeem, Dr. Sarah Nadeem, MD, FACE, Assistant Professor Dept of Medicine, Section of Endocrinology, Aga Khan University
Other Study IDs: 2020-5368-14553
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Career Choice of Medicine
Keywords: Medical education; Pre-Medical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention was done.

SUMMARY:
The aim of this study is to determine what impact the COVID-19 pandemic may have had on the choices of high school students to pursue medicine as a career.

DETAILED DESCRIPTION:
The COVID-19 pandemic poses an unprecedented global health crisis that has affected healthcare systems around the world. Those working in the health sector are at the forefront of this pandemic and naturally have been deeply impacted by it. Health care workers are at risk of serious physical exhaustion owing to long shifts, a major increase in workload and working under high-stress conditions. Shortage of Personal Protective Equipment (PPE) in many hospitals carries a serious health risk for not only healthcare workers but their families and patients as well. In addition to the physical toll that the pandemic has taken on doctors and other healthcare professionals, it has also affected their mental health deeply with an increase in anxiety and depression. Witnessing firsthand what this virus can do, yet stepping in daily into a high-risk area and exposing oneself to possible risk of infection, takes its toll on one's psychological well-being. However, the pandemic has allowed health care professionals to show higher levels of perseverance and professionalism in the face of the pandemic.

In view of how the COVID-19 pandemic has affected healthcare workers and the perception of the medical field around the world, the aim of this cross-sectional study is to determine what impact this may have had on the choices of high school students to pursue medicine as a career.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years old and ≤ 20 years old
* Enrolled in a high school in Pakistan for the academic year 2019-2020
* Can communicate in English

Exclusion Criteria:

- Studying a humanities, commerce, or pre-engineering track in high school

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pakistani high school students
Sampling Method: Non-Probability Sample
Enrollment: 1695 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
The change in the percentage (%) of students considering a career in medicine before the COVID-19 pandemic vs. after onset of the COVID-19 pandemic | 1 year
  This outcome would be measured by a self-designed questionnaire via a dichotomous question

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Nadeem, MD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No